CLINICAL TRIAL: NCT06068634
Title: Patient-Centered Care Survey of Infertility Patients
Brief Title: Patient-Centered Care Survey
Acronym: PCCS
Status: Completed | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: FER-CSS-2023-0248
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Infertility
Keywords: Patient-centered care; Patient experience
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Current Patients: Current patient is defined as any patient who has had any type of visit at a participating clinic within the last 6 months of the date of study initiation.

SUMMARY:
The key to patient-centered care is to identify what the patient perceives as meaningful. The primary objective of this research is to evaluate which aspects of patient-centered care are priorities to infertility patients, and if those priorities vary by geographical region.

DETAILED DESCRIPTION:
An electronic survey will be distributed to current patients within The Prelude Network, a network of fertility practices, for a total of six months. Survey responses will be collected anonymously using Survey Monkey. The survey is designed to collect information on patient preferences for patient-centered care. Participants will rank the importance of the different options within each Factor category (Clinic, Physician, Finance, and Staff). In addition, demographic questions are included and will be utilized to determine if these factors could have a significant impact on patient-centered care preferences. It is anticipated that at least 1,000 completed surveys will be collected. A similar survey was distributed to Prelude Network physicians. Patient and physician responses may be compared as part of additional data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Current patient within The Prelude Network (a network of fertility clinics).
* Has had any type of visit at a participating clinic within the last 6 months of the date of study initiation.

Exclusion Criteria:

* Not a current patient at a participating clinic.
* Has not had an appointment within 6 months of the date of study initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertility patients who have had any type of visit at a participating clinic within the last 6 months of the date of study initiation. Participating clinics are United States based fertility clinics who are part of The Prelude Network. This includes 10 fertility practices, consisting of approximately 40 individual locations.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Descriptive Analysis | 6 months
  Descriptive analyses of survey results.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Domar, PhD, Principal Investigator — Inception Fertility
Locations (1):
- Inception Fertility, LLC, Houston, Texas, United States

REFERENCES:
- [Background] Chen TH, Chang SP, Tsai CF, Juang KD. Prevalence of depressive and anxiety disorders in an assisted reproductive technique clinic. Hum Reprod. 2004 Oct;19(10):2313-8. doi: 10.1093/humrep/deh414. Epub 2004 Jul 8. PMID 15242992
- [Background] den Breejen EM, Nelen WL, Schol SF, Kremer JA, Hermens RP. Development of guideline-based indicators for patient-centredness in fertility care: what patients add. Hum Reprod. 2013 Apr;28(4):987-96. doi: 10.1093/humrep/det010. Epub 2013 Feb 14. PMID 23411619
- [Background] Domar AD, Gross J, Rooney K, Boivin J. Exploratory randomized trial on the effect of a brief psychological intervention on emotions, quality of life, discontinuation, and pregnancy rates in in vitro fertilization patients. Fertil Steril. 2015 Aug;104(2):440-51.e7. doi: 10.1016/j.fertnstert.2015.05.009. Epub 2015 Jun 13. PMID 26072382
- [Background] Domar AD, Rooney K, Hacker MR, Sakkas D, Dodge LE. Burden of care is the primary reason why insured women terminate in vitro fertilization treatment. Fertil Steril. 2018 Jun;109(6):1121-1126. doi: 10.1016/j.fertnstert.2018.02.130. PMID 29935647
- [Background] Garcia D, Bautista O, Venereo L, Coll O, Vassena R, Vernaeve V. Training in empathic skills improves the patient-physician relationship during the first consultation in a fertility clinic. Fertil Steril. 2013 Apr;99(5):1413-1418.e1. doi: 10.1016/j.fertnstert.2012.12.012. Epub 2013 Jan 5. PMID 23294674
- [Background] Huppelschoten AG, Aarts JW, van Empel IW, Cohlen BJ, Kremer JA, Nelen WL. Feedback to professionals on patient-centered fertility care is insufficient for improvement: a mixed-method study. Fertil Steril. 2013 Apr;99(5):1419-27. doi: 10.1016/j.fertnstert.2012.12.024. Epub 2013 Jan 26. PMID 23357454
- [Background] Pasch LA, Holley SR, Bleil ME, Shehab D, Katz PP, Adler NE. Addressing the needs of fertility treatment patients and their partners: are they informed of and do they receive mental health services? Fertil Steril. 2016 Jul;106(1):209-215.e2. doi: 10.1016/j.fertnstert.2016.03.006. Epub 2016 Mar 24. PMID 27018159
- [Background] Troude P, Ancelet S, Guibert J, Pouly JL, Bouyer J, de La Rochebrochard E. Joint modeling of success and treatment discontinuation in in vitro fertilization programs: a retrospective cohort study. BMC Pregnancy Childbirth. 2012 Aug 3;12:77. doi: 10.1186/1471-2393-12-77. PMID 22862824
- [Background] Troude P, Guibert J, Bouyer J, de La Rochebrochard E; DAIFI Group. Medical factors associated with early IVF discontinuation. Reprod Biomed Online. 2014 Mar;28(3):321-9. doi: 10.1016/j.rbmo.2013.10.018. Epub 2013 Oct 31. PMID 24461478
- [Background] van Empel IW, Dancet EA, Koolman XH, Nelen WL, Stolk EA, Sermeus W, D'Hooghe TM, Kremer JA. Physicians underestimate the importance of patient-centredness to patients: a discrete choice experiment in fertility care. Hum Reprod. 2011 Mar;26(3):584-93. doi: 10.1093/humrep/deq389. Epub 2011 Jan 12. PMID 21227936